CLINICAL TRIAL: NCT04571294
Title: Para-aortic Lymphnodes Removal During Upfront Pancreaticoduodenectomy for Pancreatic Ductal Adenocarcinoa: Should it be Performed? A Multicentre Randomized Controlled Trial.
Brief Title: Para-aortic Lymphnodes Removal During Upfront Pancreaticoduodenectomy
Acronym: PALN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Alessandro Zerbi, Professor of Surgery, Humanitas Hospital, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 451/20
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pancreas Cancer; Pancreaticoduodenal Lymphadenopathy; Pancreas Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): PALN removal
  Interventions: Procedure: removal of para-aortic lymphnodes (PALN)
- group B (No Intervention): No PALN removal

INTERVENTIONS:
Procedure: removal of para-aortic lymphnodes (PALN) — During pancreaticoduodenectomy, para-aortic lymphnodes (PALN) will be removed for the surgeon
  Arms: group A

SUMMARY:
Pancreaticoduodenectomy (PD) associated with lymphadenectomy is the only curative option for patients affected by pancreatic ductal adenocarcinoma (PDAC). In 2014, the International Study Group on Pancreatic Surgery (ISGPS) defined the "standard lymphadenectomy", that is mandatory during PD for PDAC. Lymphadenectomy should include the removal of the hepatoduodenal ligament nodes (stations 5, 6, 12b1, 12b2, 12c according the classification of Japanese Pancreas Society), nodes along the hepatic artery (station 8a), the posterior surface of the pancreatic head (station 13a and 13b), the superior mesenteric artery (14a right lateral side, 14b right lateral side) and nodes of the anterior surface of the pancreatic head (stations 17a and 17b). The inclusion of para-aortic lymphnodes (PALN) (station 16) in standard lymphadenectomy is still matter of debate. Moreover, some retrospectives or prospective studies reported that the presence of PALN metastases has a significant negative prognostic impact. Until now, no randomized studies comparing PD associated with standard lymphadenectomy with or without removal of PALN have been published. The aim of this study is to evaluate if the removal of station 16 should be routinely included in standard lymphadenectomy during PD for PDAC.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) with lymphadenectomy is the current treatment of pancreatic ductal adenocarcinoma (PDAC). The optimal lymphadenectomy during PD (standard versus extended) has been largely debated during the last two decades. Four randomized controlled trials (RCTs) published afterward reported no survival benefit, and no arguments could be presented based on the evidence of these studies to support the role of extended lymphadenectomy during PD. A similar conclusion was underlined also in two meta-analyses, the first from Michalski et al., in which 3 RCTs were analyzed, and the second from Iqbal et al., in which both RCTs and cohort studies were included, both of which showed no benefit of extended lymphadenectomy. However, the definition of lymphadenectomy varied considerably between the RCTs. For this reason, in 2014, the International Study Group on Pancreatic Surgery (ISGPS) defined the "standard lymphadenectomy" during PD for PDAC. Lymphadenectomy should include the removal of the hepatoduodenal ligament nodes (stations 5, 6, 12b1, 12b2, 12c according the classification of Japanese Pancreas Society), nodes along the hepatic artery (station 8a), the posterior surface of the pancreatic head (station 13a and 13b), the superior mesenteric artery (14a right lateral side, 14b left lateral side) and nodes of the anterior surface of the pancreatic head (stations 17a and 17b). Para-aortic lymph nodes (PALN; station 16) are considered as "extra-regional" lymph nodes. Some questions about PALN still remain open: a) should the removal of station 16 be routinely included in the standard lymphadenectomy during PD for PDAC? b) in case of removal of station 16 and intraoperative demonstration of PALN metastases at frozen section, should PD be avoided ? Several retrospective reports described that the prognosis of patients with metastatic PALN is significantly worse if compared with patients with negative PALN. Two recent-metaanalyses have been published on this topic, confirming that PALN metastases correlated with poor prognosis in patients with PDAC. However, these meta-analyses concluded that, due to the presence of some long survivors even in cases of PALN metastases, the definitive avoidance of PD in these cases needs further investigation. Until now, no consensus in case of intraoperative metastatic PALN has been reached. Moreover, it's not still clear if the removal of PALN during PD should be routinely performed. Until now, no randomized studies comparing PD with or without removal of PALN have been published. In 2014, during the consensus meeting of ISGPS, there was extensive discussion about PALN removal: no strong recommendation was formulated on dissecting station 16 routinely and it was not included in standard lymphadenectomy. For this reason, we decided to plan this multicentric RCT that compares upfront PD with and without the removal of PALN, in order to evaluate if their removal should be routinely included in standard lymphadenectomy during PD for PDAC.

ELIGIBILITY:
Inclusion Criteria:

* pre-operative radiological or histological diagnosis of pancreatic head PDAC, including PDAC arising from IPMN (invasive-IPMN) (in case of not confirmation of PDAC at final pathological examination, the case will be considered as a "drop out" and excluded from the study);
* upfront PD associated with standard lymphadenectomy.

Exclusion Criteria:

* PD performed after neoadjuvant treatment;
* PALN metastases diagnosed by a pre-operative PET-FDG (if performed);
* intraoperative distant metastases;
* R2 resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 48 months
  The primary endpoint is to compare overall survival (OS) in patients with (group A) and without (group B) removal of PALN

SECONDARY OUTCOMES:
PALN metastases | 12 months
  to evaluate the rate of PALN metastases (for group A, only)
DFS in case of PALN metastases | 48 months
  to evaluate the prognostic impact, in terms of Disease Free Survival (DFS), of PALN metastases (for group A, only)
OS in case of PALN metastases | 48 months
  to evaluate the prognostic impact, in terms of OS, of PALN metastases (for group A, only)
predictive factors of PALN metastases | 12 months
  to evaluate possible pre- and intra-operative predictive factors of PALN metastases (for group A, only)
overall post-operative morbidity | 12 months
  to compare overall post-operative morbidity rate in both study groups
post-operative pancreatic fistula (POPF) | 12 months
  to compare the POPF rate in both study groups
post-operative pancreatic haemorrhage (PPH) | 12 months
  to compare the rate of PPH in both groups
90-day mortality | 12 months
  to compare the 90-day mortality rate in both study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy/Milan, Italy